CLINICAL TRIAL: NCT03201666
Title: Comparison of Karyotyping, CMA and NIPT for Prenatal Diagnosing Chromosomal Anomalies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: YiYang Zhu (Other)
Responsible Party: Sponsor-Investigator, YiYang Zhu, Director,Clinical dean of Prenatal Diagnosis Center, Taizhou Hospital
Organization: Taizhou Hospital (Other)
Other Study IDs: TZ201607
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Prenatal Diagnosis
Keywords: prenatal diagnosis; non-invasive prenatal tests; chromosome microarray analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sample1.maternal peripheral blood，which used for extracted fetal free DNA for NIPT examination Sample2.amniotic fluid, which used for karyotyping and CMA analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This diagnostic test is aimed to compare the Karyotyping, CMA and NIPT for prenatal diagnosing chromosomal anomalies. Pregnant women who needed prenatal genetic diagnosis meted the study criterion; fetal amniotic fluid was regular examined by Karyotyping and CMA, and maternal peripheral blood was collected for NIPT detecting. And the CMA result as a golden standard, the main outcome is compared the diagnostic efficacy of NIPT for diagnosing chromosomal anomalies.

DETAILED DESCRIPTION:
Aim: to compare the Karyotyping, CMA and NIPT for prenatal diagnosing chromosomal anomalies.

Design: diagnostic test Set: Prenatal diagnosis center of Taizhou City Study population: The Pregnant women who needed amniocenteses for prenatal genetic diagnosis were recruited.

Methods: amniotic fluid was regular examined by Karyotyping and CMA, and maternal peripheral blood was used for collected for NIPT detecting.

Statistic: CMA result as a golden standard, the main outcome is compared the diagnostic efficacy of NIPT for diagnosing chromosomal anomalies.

ELIGIBILITY:
Inclusion Criteria:

1. pregnant women who needed amniocenteses were recruited during the study period, include high risk for serum screening, aged over 35 years and ultrasound abnormal.
2. only singleton were included

Exclusion Criteria:

1. women who met the contraindication for invasive procedure as : threaten abortion, acute infectious disease.
2. Women who unfitted for NIPT analysis include multiple, history of allogeneic blood cell transfusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pregnant women who needed amniocenteses were recruited during the study period
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-07-01 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
accuracy of NIPT for prenatal diagnosing chromosomal anomalies | July,2016-July, 2017
  sensitive, false negative rate, and false positive rate of NIPT compared with CMA

CONTACTS AND LOCATIONS:
Overall Officials: YiYang Zhu, MD, Study Director — prenatal doagnosis center of taizhou city
Locations (1):
- Taizhou Hospital of Zhejiang province, Taizhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No